CLINICAL TRIAL: NCT00741182
Title: Effect of PTH(1-34) Treatment on Fracture Healing in Vivo
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: The Danish Medical Research Council (Other)
Responsible Party: Peter Schwarz, Professor, MD, DMSci, Glostrup University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAO_06_011; EudraCT 2008-000094-37
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2009-08

CONDITIONS: Shoulder Fractures; Trochanteric Fractures
Keywords: Fracture; Osteoporosis; Forsteo; Teriparatide; Fracture healing
MeSH Terms: conditions — Shoulder Fractures; Hip Fractures; Fractures, Bone; Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Femur PTH(1-34) (Experimental): 24 participants with trochanteric fractures will be assigned to Forsteo (PTH(1-34)) treatment
  Interventions: Drug: rhPTH(1-34)
- Femur Control (No Intervention): 24 participants with trochanteric fractures will be assigned to "no treatment"
- Humerus PTH(1-34) (Experimental): 24 participants with collum chirurgicum fracture will be assigned to Forsteo (PTH(1-34)) treatment
  Interventions: Drug: rhPTH(1-34)
- Humerus Control (No Intervention): 24 participants with collum chirurgicum fracture will be assigned to "no treatment".

INTERVENTIONS:
Drug: rhPTH(1-34) — Injection of 20 micrograms per day in eight weeks
  Other Names: Forsteo; Forteo; Teriparatide
  Arms: Femur PTH(1-34); Humerus PTH(1-34)

SUMMARY:
The purpose of the study is to investigate, whether PTH(1-34) is able to promote fracture healing in postmenopausal women with fractures of the hip or shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Acute new osteoporotic trochanteric or collum chirurgicum fracture
* Postmenopause

Exclusion Criteria:

* Calcium metabolic disease other than osteoporosis
* Diseases known to affect calcium homeostasis
* Dementia
* Hypersensitivity to drug or other components of medication
* pre-existing hypercalcemia
* Decreased kidney function
* Increased alkaline phosphatase
* Prior external radiation therapy or brachytherapy of the skeleton
* Skeletal malignancies or bone metastases
* Alcohol and/or drug abuse
* Systemic treatment with corticosteroids within the last four weeks
* Non-cooperating patients
* Patients who do not speak and understand the danish language

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Radiological evaluation of healing | 0, 4, 8, 12, (16) weeks after fracture

SECONDARY OUTCOMES:
Biochemical bone markers | 0, 1, 2, 3, 4, 8, 12, (16) weeks after fracture
SF-36 questionnaire | 0, 4, 8, 12, (16) weeks after fracture

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schwarz, MD, DMSci, Principal Investigator — Glostrup University Hospital
Locations (1):
- Research Center for Ageing and Osteoporosis, Glostrup University Hospital, Copenhagen, Denmark